CLINICAL TRIAL: NCT04402762
Title: Pharmacodynamic Equivalence of Ovine Enoxaparin to Porcine Enoxaparin (Lovenox®) in Healthy Volunteers
Brief Title: Pharmacodynamic Equivalence of Ovine Enoxaparin to Lovenox®
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: PT Metiska Farma (Unknown)
Responsible Party: Principal Investigator, Prof. Arini Setiawati, PhD, Prof, PhD, Indonesia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CRSU.P.Enox/06.01/11/19
Record Dates: First submitted 2020-04-09; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Enoxaparin
Keywords: pharmacodynamic equivalence; anticoagulant; antithrombotic
MeSH Terms: interventions — Enoxaparin

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, 2-way cross-over, single-dose study with at least 7 days wash-out period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR treatment sequence (Experimental): Period 1-Test Treatment: Ovine enoxaparin sodium 60 mg SC injection, manufactured by Metiska Farma. Period 2-Reference Treatment: Porcine enoxaparin sodium 60 mg SC injection (Lovenox), manufactured by Sanofi, France.
  Interventions: Drug: Ovine Enoxaparin; Drug: Enoxaparin Prefilled Syringe [Lovenox]
- RT treatment sequence (Active Comparator): Period 2-Reference Treatment: Porcine enoxaparin sodium 60 mg SC injection (Lovenox), manufactured by Sanofi, France. Period 1-Test Treatment: Ovine enoxaparin sodium 60 mg SC injection, manufactured by Metiska Farma.
  Interventions: Drug: Ovine Enoxaparin; Drug: Enoxaparin Prefilled Syringe [Lovenox]

INTERVENTIONS:
Drug: Ovine Enoxaparin — The test drug is ovine enoxaparin sodium 60 mg (0.6 mL taken from 1.0 mL vial containing 100 mg = 10,000 IU anti-FXa), from Metiska Farma.
  Other Names: Ovine Enoxaparin Sodium; Ovine Enoxaparin (Metiska Farma)
Drug: Enoxaparin Prefilled Syringe [Lovenox] — The reference drug is enoxaparin sodium 60 mg (Lovenox® 0.6 mL prefilled syringe containing 60 mg = 6,000 IU anti-FXa) from Sanofi, France.
  Other Names: Active comparator

SUMMARY:
This study is designed as a randomized, open-label, 2-way cross-over, single dose study with at least 7 days wash-out period. The objective of this study is to demonstrate the pharmacodynamic / pharmacokinetic equivalence of ovine enoxaparin to the reference product, the originator porcine enoxaparin, Lovenox® from Sanofi, and to assess its safety and tolerability in healthy volunteers.

DETAILED DESCRIPTION:
Low molecular-weight heparins (LMWHs) are derived from unfractionated heparin (UFH) by chemical or enzymatic depolymerization. Enoxaparin is one of the most widely used LMWHs and is obtained by alkaline depolymerization of heparin benzyl ester derived from porcine intestinal mucosa. In contrast to UFH, enoxaparin has higher and more consistent bioavailability after s.c. administration compared with UFH and has longer plasma half-life.

Because of difficulties in chemical detection of LMWH, conventional pharmacokinetic studies cannot be performed. LMWH absorption and elimination are studied using pharmacodynamic surrogate markers, i.e. anti-FXa activity. Measurement of this pharmacodynamic activities is used to compare the biosimilar/ generic products to the reference LMWH.

This study is designed as a randomized, open-label, 2-way cross-over, single dose study with at least 7 days wash-out period. The objective of this study is to demonstrate the pharmacodynamic / pharmacokinetic equivalence of ovine enoxaparin to the reference product, the originator porcine enoxaparin, Lovenox® from Sanofi, and to assess its safety and tolerability in healthy volunteers.

The test drug is ovine enoxaparin sodium 60 mg (0.6 mL taken from 1.0 mL vial containing 100 mg = 10,000 IU anti-FXa), from Metiska Farma. Meanwhile, the reference drug is enoxaparin sodium 60 mg (Lovenox® 0.6 mL prefilled syringe containing 60 mg = 6,000 IU anti-FXa) from Sanofi, France. The drugs are not similar in appearance: ovine enoxaparin is supplied in vials, whereas Lovenox® is supplied as pre-filled syringes, both are given as s.c. injection. An unblinded pharmacist will prepare the study drug, and an unblinded medical doctor will inject the study drug.

Study procedures

1. On day-1 of period 1, subjects will be given in fasting condition, a single s.c. injection of the test or the reference drug.
2. Blood samples to assess PD parameters will be collected in both study periods at the following time points: pre-dose, and 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 16, 20, and 24 hours after dosing on Day-1 (16 sampling points).
3. Nine (9) mL of blood will be drawn from vena cubiti with a needle of 19 to 21 gauge with a maximum of 1 minute pressure with tourniquet, the first 3 mL of blood will be collected in an empty tube (to be thrown away), the second 3 mL of blood will be collected in a blood collection tube containing citrate, theophylline, adenosine, and dipyridamole (CTAD tube) for anti-FXa and anti-FIIa, and the third 3 mL of blood will be collected in a citrate tube for TFPI. In case of failure in blood drawing, the phlebotomist should change the site of blood drawing and change the needle used.
4. Subjects will return to the clinic after a wash-out period of at least 7 days, and on day-1 of period 2, they will be crossed over to receive a single s.c. dose of the alternate drug.

Anti-FXa activity will be determined by a chromogenic method using a commercial kit (STA-Liquid anti-FXa, Diagnostica Stago S.A.S, France) within 4 hours after sample collection at room temperature. Meanwhile, anti-FIIa activity will be measured by a chromogenic method using a commercial kit (Biophen anti-FIIa, STA Compact Max, France) within 4 hours after sample collection at room temperature, and TFPI levels will be measured using a commercial ELISA kit (Abcam PLC, Cambridge, UK).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers of both sexes aged 18 - 45 years with BMI 18 - 25 kg/m2 inclusive.
2. Have no clinically significant abnormalities based on medical history, clinical laboratory tests, vital sign measurements, 12-lead ECG results, and physical examination findings.
3. Willing to participate in the study by signing the informed consent.

Exclusion Criteria:

1. Female < 45 kg or male < 57 kg
2. Calculated (Cockroft & Gault formula) ClCr < 80 mL/min
3. History of or positive test result for alcohol abuse or drug addiction.
4. History of relevant drug and/or food allergies.
5. Any prescription drug (especially antiplatelet or anticoagulant drug) or OTC medication including herbal, supplement, etc. that could affect coagulation within 2 weeks before study dosing.
6. Administration of any investigational drug within 60 days before study drug dosing.
7. Taking anti TB rifampicin within 60 days before study drug dosing.
8. A positive test for HIV (1 or 2) Ab, HBsAg, or HepC Ab.
9. A positive fecal occult blood at screening.
10. History and/or current conditions of bleeding tendency.
11. History of thrombocytopenia, including heparin-induced (by anamnesis).
12. Known history of hypersensitivity to drugs with a chemical structure similar to enoxaparin sodium (eg. UFH, LMWH) or to pork or lamb products.
13. Females: - during menstruation period

    * Pregnancy or lactation
    * taking hormonal contraception (oral or injection)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-05-03 (Actual)

PRIMARY OUTCOMES:
Maximum activity (Amax) | Day -1 (periode 1 and 2), before dosing (pre-dose), and between 1 and 24 hours after dosing on day 1 (period 1 and 2)
  Amax will be measured for anti-FXa activity, anti-FIIa activity and TFPI levels
Area under the effect curve (AUEC0-t) | Day -1 (periode 1 and 2), before dosing (pre-dose), and between 1 and 24 hours after dosing on day 1 (period 1 and 2)
  The AUEC will be measured from time 0 to the last measured activity (AUEC0-t) of anti-FXa activity, anti-FIIa activity, and TFPI levels

SECONDARY OUTCOMES:
Adverse events | From informed consent signature until the study end
  Adverse Events - total and related (ADRs) and Serious Adverse Events - total and related (SADRs)

CONTACTS AND LOCATIONS:
Overall Officials: Arini Setiawati, Prof, PhD, Principal Investigator — Clinical Research Supporting Unit, Faculty of Medicine, University of Indonesia
Locations (1):
- Pharma Metric Labs, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee S, Raw A, Yu L, Lionberger R, Ya N, Verthelyi D, Rosenberg A, Kozlowski S, Webber K, Woodcock J. Scientific considerations in the review and approval of generic enoxaparin in the United States. Nat Biotechnol. 2013 Mar;31(3):220-6. doi: 10.1038/nbt.2528. PMID 23471071
- [Result] Martinez Gonzalez J, Monreal M, Ayani Almagia I, Llaudo Garin J, Ochoa Diaz de Monasterioguren L, Gutierro Aduriz I. Bioequivalence of a biosimilar enoxaparin sodium to Clexane(R) after single 100 mg subcutaneous dose: results of a randomized, double-blind, crossover study in healthy volunteers. Drug Des Devel Ther. 2018 Mar 19;12:575-582. doi: 10.2147/DDDT.S162817. eCollection 2018. PMID 29593380
- See also: EMA Assessment report for Inhixa (enoxaparin sodium), 2016 — https://www.ema.europa.eu/en/documents/assessment-report/inhixa-epar-public-assessment-report_en.pdf